CLINICAL TRIAL: NCT03784612
Title: The HAPPY-study: Digital Support for Healthier Eating Habits in Patients with Diabetes Type 2 - a Randomized Clinical Trial Within Primary Care
Brief Title: The Healthy Eating with APP TechnologY Study
Acronym: HAPPY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Stephanie Bonn, PhD, Assistant professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Dnr: 2018/652-31
Record Dates: First submitted 2018-12-14; First posted 2018-12-24 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2023-10

CONDITIONS: Type 2 Diabetes Mellitus; Dietary Habits
Keywords: Smartphone application; HbA1c; Blood lipids; Dietary intake
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- App-technology group (Experimental): Participants in the App-technology group arm will use a newly developed smartphone application ("app"), containing a 12-week healthy eating program.
  Intervention: App-technology for healthy eating habits.
  Interventions: Behavioral: App-technology for healthy eating habits
- Control group (No Intervention): The control group will receive standard care.

INTERVENTIONS:
Behavioral: App-technology for healthy eating habits — Access to smartphone-app, including a 12 week healthy eating program. A new theme on healthy dietary habits is presented each week.
  Arms: App-technology group

SUMMARY:
The aim of this study is to investigate the effect of using new app-based technology to improve dietary habits, compared to usual care in patients with type 2 diabetes. The hypothesis is that the intervention, i.e. using the new technology an an app-based course for healthy eating habits, will have a greater positive effect on dietary habits and biological markers, including HbA1c and serum lipids, than usual care.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of type 2 diabetes
* 18 years of age or older
* Ability to communicate in Swedish
* Own and use a smartphone with a personal digital ID

Exclusion criteria:

- No specific exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Change in dietary intake | Baseline and month 3, and 6
  Change in dietary intake assessed using a four day food record.

SECONDARY OUTCOMES:
HbA1c | Baseline and month 3, and 6
  mmol/mol, Heamoglobin A1c
Total cholesterol | Baseline and month 3, and 6
  mmol/L
HDL-cholesterol | Baseline and month 3, and 6
  mmol/L
Triglycerides | Baseline and month 3, and 6
  mmol/L
Body Mass Index (BMI) | Baseline and month 3, and 6
  kg/m2, measured height and weight
Body weight | Baseline and month 3, and 6
  kg, measured
Body composition: Body fat | Baseline and month 3, and 6
  Body fat (kg), measured using a bioelectrical scale
Body composition: Fat free mass | Baseline and month 3, and 6
  Fat free mass (kg), measured using a bioelectrical scale
Body composition: Muscle mass | Baseline and month 3, and 6
  Muscle mass (kg), measured using a bioelectrical scale
Body composition: Total body water | Baseline and month 3, and 6
  Total body water (kg), measured using a bioelectrical scale
Waist circumference | Baseline and month 3, and 6
  cm, measured
Blood pressure | Baseline and month 3, and 6
  mmHg, measured

OTHER OUTCOMES:
Change in dietary intake and eating habits | Baseline and month 3, 6 and 12
  Assessed using a 94 item food frequency questionnaire (FFQ)
Change in eating behaviour assessed using Three-Factor Eating Questionnaire-R21 (TFEQ-R21) | Baseline and month 3, 6 and 12
  Assessed using a 21-item questionnaire
Change in physical activity assessed using the Active-Q questionnaire | Baseline and month 3, 6 and 12
  Assessed using a 48 item questionnaire including activities in domains of Daily occupation, transportation, leisure time, and exercise
Change in self-reported medication use | Baseline and month 3, 6 and 12
  One question on medication use for blood sugar levels and one questions on medication use for blood lipid levels
Change in tobacco use habits | Baseline and month 3, 6 and 12
  Two questions regarding smoking and Swedish snuff use
Change in sleeping habits | Baseline and month 3, 6 and 12
  Assessed using a modified 13-item Karolinska Sleep questionnaire
Change in perceived purpose in Life (PIL) | Baseline and month 3, 6 and 12
  Assessed using 6-item questionnaire
Change in perceived stress levels | Baseline and month 3, 6 and 12
  Assessed using the 14-item perceived stress scale (PSS)
Change in self-reported diabetes self-efficacy | Baseline and month 3, 6 and 12
  Assessed using a 20-item questionnaire
Change in health related quality of life | Baseline and month 3, 6 and 12
  Assessed using the 36-item RAND-36 questionnaire
Change in perceived social support from family and friends for healthy eating habits | Baseline and month 3, 6 and 12
  Assessed using a 3-item questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie E Bonn, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cecchini V, Sjoblom L, Lagerros YT, Bonn SE. The Effect of a Mobile Health Dietary Education Intervention on Ultra-processed Food Consumption in Patients with Type 2 Diabetes: A Randomized Controlled Trial. Curr Dev Nutr. 2025 Apr 28;9(6):107454. doi: 10.1016/j.cdnut.2025.107454. eCollection 2025 Jun. PMID 40510749
- [Derived] Sjoblom L, Hantikainen E, Dahlgren A, Trolle Lagerros Y, Bonn SE. The effect of an app-based dietary education on dietary intake and cardiometabolic risk markers in people with type 2 diabetes: results from a randomized controlled trial. Nutr J. 2025 Jan 4;24(1):2. doi: 10.1186/s12937-024-01069-2. PMID 39754157
- [Derived] Pitt S, Sjoblom L, Balter K, Trolle Lagerros Y, Bonn SE. The effect of an app-based dietary intervention on diet-related greenhouse gas emissions - results from a randomized controlled trial. Int J Behav Nutr Phys Act. 2023 Oct 11;20(1):123. doi: 10.1186/s12966-023-01523-0. PMID 37821876
- [Derived] Trolle Lagerros Y, Dahlgren A, Sjoblom L, Bonn SE. Digital Support for Healthier Eating Habits Among Patients With Type 2 Diabetes: Protocol for a Randomized Clinical Trial Within Primary Care (HAPPY Trial). JMIR Res Protoc. 2020 Nov 16;9(11):e24422. doi: 10.2196/24422. PMID 33196448